CLINICAL TRIAL: NCT02918292
Title: Optimizing Haploidentical Aplastic Anemia Transplantation (CHAMP) (BMT CTN 1502)
Brief Title: Optimizing Haploidentical Aplastic Anemia Transplantation (BMT CTN 1502)
Acronym: CHAMP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT CTN 1502; 2U10HL069294-11 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Results first posted 2022-07-12 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Severe Aplastic Anemia
Keywords: Haploidentical Bone Marrow; Hematopoietic Stem Cell Transplant (HSCT); Severe Aplastic Anemia (SAA); Antithymocyte Globulin (ATG)
MeSH Terms: conditions — Anemia, Aplastic | interventions — Antilymphocyte Serum; thymoglobulin; fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Haplo Bone Marrow HSCT (Experimental): Patients will be treated with a preparative regimen of Antithymocyte Globulin (ATG) (4.5 mg/kg), fludarabine (150 mg/m^2), cyclophosphamide (29 mg/kg), and low dose total body irradiation (TBI) (200 cGy) before undergoing the haplo HSCT. GVHD prophylaxis will be with post-HSCT cyclophosphamide (100 mg/kg), tacrolimus, and mycophenolate mofetil (MMF). G-CSF will be administered post-transplant.
  Interventions: Drug: Antithymocyte Globulin (ATG); Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation (TBI); Procedure: Haplo HSCT; Drug: Tacrolimus; Drug: Mycophenolate mofetil (MMF); Drug: G-CSF

INTERVENTIONS:
Drug: Antithymocyte Globulin (ATG) — Administration of ATG will be 0.5 mg/kg IV on Day -9 over 6 hours and 2 mg/kg IV on Days -8 and -7 over 4 hours.
  Other Names: Thymoglobulin®, rATG
Drug: Fludarabine — Fludarabine dose will be 30 mg/m^2 IV daily for 5 days from Day -6 to Day -2.
  Other Names: Fludara®
Drug: Cyclophosphamide — Cyclophosphamide dose will be 14.5 mg/kg IV daily for 2 days (Day -6 to Day -5) prior to transplantation and 50 mg/kg IV daily for 2 days (Day +3 to Day +4) after transplantation.
  Other Names: Cytoxan®
Radiation: Total Body Irradiation (TBI) — TBI is to be delivered in a single dose of 200 cGy on Day -1.
Procedure: Haplo HSCT — Eligible patients without a fully matched related or unrelated donor available will undergo haploidentical bone marrow transplant.
Drug: Tacrolimus — Tacrolimus should be started on Day +5 and administered to maintain a level of 10-15 ng/mL.
  Other Names: Prograf®
Drug: Mycophenolate mofetil (MMF) — MMF dose will be 15 mg/kg PO three times a day (TID) up to 1 gm TID (or IV equivalent) starting on Day +5.
  Other Names: Cellcept®
Drug: G-CSF — G-CSF will be given IV or SQ starting on Day +5 at 5 mcg/kg/day until ANC is > 1500 for 3 days.
  Other Names: Filgrastim, Neupogen®

SUMMARY:
This study is a prospective, multicenter phase II study with patients receiving haploidentical transplantation for Severe Aplastic Anemia (SAA). The primary objective is to assess overall survival (OS) at 1 year post-hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
Acquired SAA is a rare bone marrow failure disorder with an estimated annual incidence of 2 cases per million and with over 600 new cases in the United States each year. A major challenge in treating acquired SAA is the management of patients who are refractory to immunosuppressant therapy (IST) or have relapsed after IST. HSCT is the only curative option for these patients but many are ineligible because they lack a suitable donor. The Blood and Marrow Transplant Clinical Trials Network (BMT CTN) seeks to increase options for these patients by using novel therapeutic strategies of GVHD prophylaxis with PTCy to expand the donor pool to include haploidentical donors. The goal of this protocol is to test whether optimized approaches using haploidentical donors will achieve acceptable outcomes in SAA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is < 75 years of age at time of enrollment.
2. Confirmed diagnosis of SAA, either from initial diagnosis or follow-up assessments, defined as:

   1. Bone marrow cellularity < 25% or marrow cellularity < 50% but with < 30% residual hematopoietic cells.
   2. Two out of three of the following (in peripheral blood): Neutrophils < 0.5 x10^9/L, Platelets < 20 x10^9/L, or Reticulocyte count < 20 x10^9/L (<60 x 10^9/L using an automated analysis)
3. No suitable fully matched related sibling donor (6/6 match for human leukocyte antigen (HLA)-A and B at intermediate or high resolution and DRB1 at high resolution using DNA-based typing) available.
4. Failed at least one trial of immunosuppressive therapy (IST) by being refractory or having relapsed. IST could have included ATG based regimens, calcineurin inhibitors and/or other higher dose therapy directed at the treatment of primary SAA.
5. Available relative of the patient who is a haploidentical match, including biological parents, siblings or half siblings, children, uncles/aunts, first cousins, etc. Eligible haploidentical donors will have 2-4 mismatches if HLA-A, -B, -C, and -DRB1 typing is used; 2-5 mismatches if HLA-A, -B, -C, -DRB1, and -DQB1 typing is used; and 2-6 mismatches if HLA-A, -B, -C, -DRB1, -DQB1, and -DPB1 typing is used. A unidirectional mismatch in either the graft versus host or host versus graft direction is considered a mismatch. The donor and recipient must demonstrate that they are a full haplotype match by being identical at a minimum of one allele (at high resolution DNA-based typing) at the following genetic loci: HLA-A, -B, -C, and DRB1 if 8 allele typing is used; HLA-A, -B, -C, -DRB1, and -DQB1 if 10 allele typing is used; and HLA-A, -B, -C, -DRB1-, DQB1, and -DPB1 is 12 allele typing is used by the local center. See Section 2.4 for additional information.
6. Patient and/or legal guardian must sign informed consent for HSCT.
7. The haplo donor and/or legal guardian must be able to sign informed consent documents.
8. The potential haplo donor must be willing and able to donate bone marrow.
9. The weight of the haplo donor must be ≥ 20 kg.
10. Adequate organ function defined as:

    1. Cardiac: Left ventricular ejection fraction (LVEF) at rest ≥ 40%. For patients aged < 13 years, shortening fraction (SF) ≥ 26% by echocardiogram or Multi Gated Acquisition Scan (MUGA) may be substituted for LVEF.
    2. Hepatic: Total bilirubin < 3.0 x the upper limit of normal (ULN) for age (patients who have been diagnosed with Gilbert's Disease are allowed to exceed this limit) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5.0 x ULN for age.
    3. Renal: For patients > 13.0 years of age at the time of enrollment: estimated creatinine clearance > 50 mL/minute (using the Cockcroft-Gault formula and actual body weight). For patients < 13.0 years of age at enrollment: Glomerular Filtration Rate (GFR) estimated by the updated Schwartz formula ≥ 90 mL/min/1.73 m2. If the estimated GFR is < 90 mL/min/1.73 m^2, then renal function must be measured by 24-hour creatinine clearance or nuclear GFR, and must be > 50 mL/min/1.73 m^2.
    4. Pulmonary: For patients > 13.0 years of age: Diffusing capacity of the lung for carbon monoxide (DLCO) (corrected/adjusted for hemoglobin) > 40% and forced expiratory volume in one second (FEV1) > 50% predicted (without administration of bronchodilator) and forced vital capacity (FVC) > 50% predicted. For patients < 13.0 years of age unable to perform pulmonary function tests (PFT) due to age or developmental ability: (1) no evidence of dyspnea at rest and (2) no need for supplemental oxygen and (3) O2 saturation > 92% on room air at sea level (with lower levels allowed at higher elevations per established center standard of care (e.g., Utah, 4,200 feet above sea level, does not give supplemental oxygen unless below 90%)).
11. Karnofsky or Lansky performance status ≥ 60%.
12. Females and males of childbearing potential must agree to practice 2 effective methods of contraception at the same time or agree to abstinence.

Exclusion Criteria:

1. Inherited bone marrow failure syndromes such as Fanconi anemia must be ruled out according to center standard.
2. Clonal cytogenetic abnormalities consistent with pre-myelodysplastic syndrome (pre-MDS) or MDS on marrow examination (e.g. Monosomy 7).
3. Presence of anti-donor HLA antibodies (positive anti-donor HLA antibody is defined as a positive cross-match test of any titer by complement-dependent cytotoxicity or flow cytometric testing or the presence of anti-donor HLA antibody to the high expression loci HLA-A, B, C, DRB1, or DPB1 with mean fluorescence intensity (MFI) > 1000 by solid phase immunoassay).
4. Prior allogeneic stem cell transplant.
5. Prior solid organ transplant.
6. Known life-threatening reaction (i.e., anaphylaxis) to Thymoglobulin® that would prohibit use for the patient as this study requires use of the Thymoglobulin® preparation of ATG.
7. Uncontrolled bacterial, viral, or fungal infection at the time of enrollment. Uncontrolled is defined as currently taking medication and with progression or no clinical improvement on adequate medical treatment.
8. Seropositive for the human immunodeficiency virus (HIV).
9. Active Hepatitis B or C determined by a detectable viral load of HBV or HCV.
10. Female patients who are pregnant (per institutional practice) or breast-feeding.
11. Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent > 5 years previously will be allowed. Cancer treated with curative intent ≤ 5 years previously will not be allowed unless approved by the Protocol Chairs and/or Protocol Officer.
12. Alemtuzumab or ATG within 2 weeks of enrollment.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research
Locations (28):
- United States (28):
  - City of Hope National Medical Center, Duarte, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Stanford Hospital and Clinics, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Gainesville, Florida
  - Miami Children's Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Indiana University Medical Center/ Riley Hospital for Children, Indianapolis, Indiana
  - University of Louisville/Kosair Children's Hospital, Louisville, Kentucky
  - Johns Hopkins Unversity, Baltimore, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute/Children's Hospital of Michigan, Detroit, Michigan
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Penn State College of Medicine/The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas/MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Children's Hospital of Wisconsin/Midwest Children's Cancer, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] DeZern AE, Eapen M, Wu J, Talano JA, Solh M, Davila Saldana BJ, Karanes C, Horwitz ME, Mallhi K, Arai S, Farhadfar N, Hexner E, Westervelt P, Antin JH, Deeg HJ, Leifer E, Brodsky RA, Logan BR, Horowitz MM, Jones RJ, Pulsipher MA. Haploidentical bone marrow transplantation in patients with relapsed or refractory severe aplastic anaemia in the USA (BMT CTN 1502): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2022 Sep;9(9):e660-e669. doi: 10.1016/S2352-3026(22)00206-X. Epub 2022 Jul 27. PMID 35907408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 14 centers between May 2017 and August 2020. The study opened to accrual on May 19, 2017 with 26 centers activated for enrollment. The study closed to accrual on August 31, 2020 and study completed on August 17, 2021. The study was initially designed to enroll participants into Unrelated Cord Blood and Haploidentical cohorts. Due to lack of accrual, the Unrelated Cord Blood cohort was closed for accrual per DSMB recommendation with no patients enrolled.
Period: Study Enrollment Prior to Transplant
Arm/Group | Haplo Bone Marrow HSCT
Started | 32
Completed | 31
Not Completed | 1
Not completed — Death | 1
Period: Study Follow up After Transplant
Arm/Group | Haplo Bone Marrow HSCT
Started | 31
Completed | 25
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes transplanted participants.
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (23.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 16
  More than one race | 1
  Unknown or Not Reported | 3
Donor age [Mean (Standard Deviation); unit: years] | 37.9 (10.8)
Donor relationship [Count of Participants; unit: Participants] — Related Haploidentical
  Participants | 31
Donor gender [Count of Participants; unit: Participants]
  Female | 18
  Male | 13
Donor Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 25
Donor Race [Count of Participants; unit: Participants]
  Asian | 4
  Black or African American | 7
  Hawaiian/Pacific Islander | 1
  White | 16
  Unknown | 3
Donor Blood Type [Count of Participants; unit: Participants]
  A+ | 10
  A- | 1
  AB+ | 1
  B+ | 6
  O+ | 9
  O- | 2
  Missing | 2
Recipient Blood Type [Count of Participants; unit: Participants]
  A+ | 8
  A- | 3
  AB+ | 3
  AB- | 1
  B+ | 5
  O+ | 10
  Missing | 1
Lansky/Karnofsky Performance Score [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    100 | 5
    90 | 13
    80 | 8
    70 | 5
Serum Bilirubin level [Mean (Standard Deviation); unit: mg/dL] | 0.8 (0.4)
Creatinine clearance level [Mean (Standard Deviation); unit: mL/min] — Creatinine clearance is estimated by using Cockcroft-Gault formula and actual body weight. Population: Serum Creatinine level is only measured for Participants >= 13.0 years old at the time of enrollment.
  mL/min
    number analyzed (Participants) | 23
    (all) | 100.9 (36.2)
Recipient-to-Donor HLA Match Scores [Count of Participants; unit: Participants] — HLA Match Score includes genetic matching information at HLA-A, -B, and -DRB1 loci or HLA-A, -B, -C, and -DRB1 loci. Matching at all HLA-A, -B, -C, and -DRB1 loci is designated as 8/8 HLA matching. A 6/8 HLA match includes mismatches at any two loci.
  Participants
    4/8 | 18
    5/8 | 8
    6/8 | 3
    7/8 | 2
TNC count [Mean (Standard Deviation); unit: x10^8 cells] — The total nucleated cells is calculated by multiplying the volume of the marrow by the marrow nucleated cell count. Prior to the procedure, determine the weight of the collection bag or tare the scale. The weight of the product (total weight minus bag or weight above the tared weight) is then divided by 1.058, the specific gravity of marrow. This result is the volume of the marrow. The marrow nucleated cell count is determined by the nucleated cell count from the lab in cells/mL corrected by subtracting the number of peripheral blood white cells/mL presumed to be contaminating the marrow.
  x10^8 cells | 204.9 (93.3)
TNC per kg Recipient Body Weight [Mean (Standard Deviation); unit: × 10^8 cells/kg] — The total nucleated cells is calculated by multiplying the volume of the marrow by the marrow nucleated cell count. Prior to the procedure, determine the weight of the collection bag or tare the scale. The weight of the product (total weight minus bag or weight above the tared weight) is then divided by 1.058, the specific gravity of marrow. This result is the volume of the marrow. The marrow nucleated cell count is determined by the nucleated cell count from the lab in cells/mL corrected by subtracting the number of peripheral blood white cells/mL presumed to be contaminating the marrow.
  × 10^8 cells/kg | 4.4 (1.7)
CD34 Count [Mean (Standard Deviation); unit: x10^6 cells] | 213.8 (139.2)
CD34 Count per kg Recipient Body Weight [Mean (Standard Deviation); unit: × 10^6 cells/kg] | 4.7 (2.7)
RBC Count [Mean (Standard Deviation); unit: million/uL] | 2.7 (0.4)
CD3 Count [Mean (Standard Deviation); unit: cells/uL] | 862.0 (631.5)
CD3 Count per kg Recipient Body Weight [Mean (Standard Deviation); unit: cells/uL per kg] | 21.9 (20.3)
Interval from Diagnosis to Transplant [Mean (Standard Deviation); unit: months] | 23.8 (26.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Survival (OS)
Description: Overall survival (OS) is the primary endpoint of this study. The time to this event is the time from transplant to death from any cause or last follow-up or 1 year from transplant, whichever occurs first. The one-year OS probability and its 95% confidence interval were estimated using the Kaplan-Meier estimator and Greenwood's formula.
Time Frame: 1 year
Population: Analysis Population includes transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
percentage of participants | 80.6 [61.9 to 90.8]

2. Secondary Outcome: Percentage of Participants With Neutrophil Recovery
Description: Neutrophil recovery is achieving an absolute neutrophil count (ANC) > 0.5 x10^9/L for three consecutive measurements on different days, with the first of the three days being defined as the day of neutrophil engraftment. The cumulative percentage of neutrophil engraftment was estimated with a 95% confidence interval using the Aalen-Johansen estimator with death prior to neutrophil engraftment treated as a competing risk.
Time Frame: Day 28 and 56
Population: Analysis Population includes transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
percentage of participants
  Day 28 | 93.5 [72.4 to 98.6]
  Day 56 | 93.5 [72.4 to 98.6]

3. Secondary Outcome: Percentage of Participants With Platelet Recovery
Description: Platelet recovery is defined by achieving a platelet count > 20 x 10^9/L with no platelet transfusions in the preceding seven days. The first day of the sustained platelet count will be defined as the day of platelet engraftment. The cumulative percentage of platelet engraftment was estimated with a 95% confidence interval using the Aalen-Johansen estimator with death prior to platelet engraftment treated as a competing risk.
Time Frame: Day 100
Population: Analysis Population includes transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
percentage of participants | 77.4 [57.3 to 88.9]

4. Secondary Outcome: Participants Alive With Sustained Engraftment
Description: Being alive and engrafted is defined as not having experienced death, primary graft failure, or secondary graft failure. Donor cell engraftment is defined as donor chimerism greater than or equal to 5% on or after Day 56 after transplantation. Chimerism may be evaluated in whole blood or blood cell fractions, including CD3 and CD33 or CD15 fractions. For this protocol, lineage-specific, myeloid, and T cell chimerisms are required. This endpoint was adjudicated by the Endpoint Review Committee (ERC) and ERC data was used for the analysis.
Time Frame: 1 year
Population: Analysis Population includes transplanted participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
Participants
  Yes, alive and engrafted | 24
  Primary graft failure | 4
  Secondary graft failure | 1
  Death without graft failure | 2

5. Secondary Outcome: Percentage of Participants With Graft-Failure-Free Survival
Description: Events for Graft-Failure-Free Survival (GFFS) including death, primary graft failure, secondary graft failure. The time to this event is the time from transplant to death from any cause, or graft failure, or last follow-up, or 1 year from transplant, whichever occurs first. For patients experiencing primary graft failure, Day 0.1 was used for primary graft failure event date to count the event in. The one-year GFFS probability and its 95% confidence interval were estimated using the Kaplan-Meier estimator and Greenwood's formula.
Time Frame: 1 year
Population: Analysis Population includes transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
percentage of participants | 77.4 [58.4 to 88.5]

6. Secondary Outcome: Percentage of Participants With Primary Graft Failure
Description: Primary graft failure is defined by the lack of neutrophil engraftment by Day 56 post-HSCT or failure to achieve at least 5% donor chimerism (whole blood or marrow) on any measurements up to and including Day +56. For this protocol, lineage-specific, myeloid, and T cell chimerisms are required. Myeloid engraftment might not proceed at the same rate as T cell engraftment. If myeloid has greater than or equal to 5% donor, even if T cell compartment does not, this is not considered primary graft failure. Secondary graft failure is defined by initial neutrophil engraftment (ANC greater than or equal to 0.5 x 10^8/L measured for 3 consecutive measurements on different days) followed by sustained subsequent decline in ANC to less than 0.5 x 10^9/L for three consecutive measurements on different days or initial whole blood or marrow donor chimerism greater than or equal to 5%, but then declining to less than 5% on subsequent measurements or second infusion/transplant given for graft failure.
Time Frame: Day 56
Population: Analysis Population includes transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
percentage of participants | 12.9 [3.6 to 29.8]

7. Secondary Outcome: Percentage of Participants With Secondary Graft Failure
Description: Secondary graft failure is defined as any one of the following:
  1. Initial neutrophil engraftment (ANC greater than or equal to 0.5 x10^9/L measured for three consecutive measurements on different days) followed by sustained subsequent decline in ANC to less than 0.5 x 10^9/L for three consecutive measurements on different days;
  2. Initial whole blood or marrow donor chimerism greater than or equal to 5%, but then declining to less than 5% on subsequent measurements;
  3. Second infusion/transplant given after Day 56 for graft failure.
Time Frame: 1 year
Population: Analysis Population includes transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
percentage of participants | 3.2 [0.1 to 16.7]

8. Secondary Outcome: Participants Alive With Autologous Recovery
Description: Autologous recovery is defined as ANC > 0.5 x 10^9/L and transfusion independence but with < 5% donor chimerism (whole blood or m. arrow). This endpoint was reviewed and adjudicated by ERC. The analysis is based on ERC data.
Time Frame: 1 year
Population: Analysis Population includes transplanted participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
Participants
  Yes, alive with autologous recovery | 0
  No, Death | 6
  No, Alive but not auto recovery | 25

9. Secondary Outcome: Percentage of Participants With Acute Graft-vs-host-disease (GVHD)
Description: Acute GVHD is graded by consensus grading (Przepiorka 1995) per BMTCTN manual of procedures (MOP). Acute GVHD is graded by consensus grading (Przepiorka 1995) per BMTCTN manual of procedures (MOP). The time of onset of grades II-IV and grades III-IV acute GVHD were recorded. This endpoint is evaluated through 100 days post-transplant. Cumulative percentage of acute GVHD post-transplant are estimated using the cumulative incidence function, treating death prior to acute GVHD as the competing risk.
Time Frame: Day 100
Population: Analysis Population includes transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
percentage of participants | 16.1 [5.7 to 31.1]

10. Secondary Outcome: Participants With Maximum Acute GVHD
Description: Acute GVHD is graded by consensus grading (Przepiorka 1995) per BMTCTN manual of procedures (MOP). Acute GVHD grading is performed by the consensus conference criteria (Przepiorka et al. 1995) with higher grade indicating worse outcomes. Grade I acute GVHD is defined as Skin stage of 1-2 and stage 0 for both GI and liver organs. Grade II is stage 3 of skin, or stage 1 of GI, or stage 1 of liver. Grade III is stage 2-4 for GI, or stage 2-3 of liver. Grade IV is stage 4 of skin, or stage 4 of liver. Maximum grade of acute GVHD through 100 days post transplant is reported.
Time Frame: Day 100
Population: Analysis Population includes transplanted participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
Participants
  None | 23
  Grade I | 3
  Grade II | 5
  Grade III | 0
  Grade IV | 0

11. Secondary Outcome: Percentage of Participants With Chronic GVHD
Description: The event for this secondary endpoint is any chronic GVHD based on 2014 NIH Consensus Criteria. This includes mild, moderate and severe chronic GVHD. The analyses of Chronic GVHD use the site-reported data. The cumulative percentage of chronic GVHD is computed using the cumulative incidence function, treating death prior to chronic GVHD as a competing risk. Eight organs will be scored on a 0-3 scale to reflect degree of chronic GVHD involvement. Liver and pulmonary function test results and use of systemic therapy for treatment of chronic GVHD will also be recorded. This secondary endpoint of chronic GVHD will include mild, moderate and severe chronic GVHD based on NIH Consensus Criteria.
Time Frame: 1 year
Population: Analysis Population includes transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
percentage of participants | 25.8 [11.9 to 42.2]

12. Secondary Outcome: Number of Participants Experiencing Chronic GVHD With Maximum Severity
Description: The event for this secondary endpoint is any chronic GVHD based on 2014 NIH Consensus Criteria. Eight organs will be scored on a 0-3 scale to reflect degree of chronic GVHD involvement. Liver and pulmonary function test results and use of systemic therapy for treatment of chronic GVHD will also be recorded. The overall chronic GVHD severity is based on the eight organs score. The maximin severity level of chronic GVHD include mild, moderate and severe.
Time Frame: 1 year
Population: Analysis Population includes transplanted participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
Participants
  None | 23
  Mild | 7
  Moderate | 1
  Severe | 0

13. Secondary Outcome: Immune Reconstitution of Flow Cytometry
Description: Quantitative assessments of peripheral blood CD3, CD4, CD8, CD19, and CD56 positive lymphocytes will be done through flow cytometric analysis.
Time Frame: Baseline, Days 100, 180, and 365
Population: Analysis Population includes transplanted participants with available data at each time point. All transplanted participants contribute data for this endpoint assessment, but not all participants provided all subsets of immune reconstitution data at each assessment time point. Only participants who had immune reconstitution results are assessed at each time point.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
cells/uL
  CD3 at Baseline: number analyzed (Participants) | 26
  CD3 at Baseline | 862 (631.5)
  CD3 at Day 100: number analyzed (Participants) | 26
  CD3 at Day 100 | 550.8 (844.1)
  CD3 at 6 Months: number analyzed (Participants) | 24
  CD3 at 6 Months | 640.5 (662.4)
  CD3 at 1 Year: number analyzed (Participants) | 21
  CD3 at 1 Year | 1121 (808.3)
  CD4 at Baseline: number analyzed (Participants) | 29
  CD4 at Baseline | 434.1 (323.3)
  CD4 at Day 100: number analyzed (Participants) | 28
  CD4 at Day 100 | 122.3 (123.1)
  CD4 at 6 Months: number analyzed (Participants) | 25
  CD4 at 6 Months | 172.6 (119.8)
  CD4 at 1 Year: number analyzed (Participants) | 22
  CD4 at 1 Year | 472.7 (365.6)
  CD8 at Baseline: number analyzed (Participants) | 26
  CD8 at Baseline | 326.9 (274.8)
  CD8 at Day 100: number analyzed (Participants) | 27
  CD8 at Day 100 | 272.9 (318.5)
  CD8 at 6 Months: number analyzed (Participants) | 23
  CD8 at 6 Months | 333.3 (409.1)
  CD8 at 1 Year: number analyzed (Participants) | 20
  CD8 at 1 Year | 569.7 (616.7)
  CD19 at Baseline: number analyzed (Participants) | 29
  CD19 at Baseline | 106.2 (159.9)
  CD19 at Day 100: number analyzed (Participants) | 28
  CD19 at Day 100 | 221.1 (477.2)
  CD19 at 6 Months: number analyzed (Participants) | 26
  CD19 at 6 Months | 204.8 (173.4)
  CD19 at 1 Year: number analyzed (Participants) | 23
  CD19 at 1 Year | 264.6 (222.3)
  CD56 at Baseline: number analyzed (Participants) | 29
  CD56 at Baseline | 124.6 (186.5)
  CD56 at Day 100: number analyzed (Participants) | 28
  CD56 at Day 100 | 237.6 (232.5)
  CD56 at 6 Months: number analyzed (Participants) | 24
  CD56 at 6 Months | 260.3 (228.6)
  CD56 at 1 Year: number analyzed (Participants) | 20
  CD56 at 1 Year | 293.2 (300.2)

14. Secondary Outcome: Immune Reconstitution of Quantitative Immunoglobulins
Description: Quantitative immunoglobulins of IgA, IgG, IgM were done at baseline and 1-year post-transplant.
Time Frame: baseline and 1-year
Population: Analysis Population includes transplanted participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
mg/dL
  IgA at Baseline | 172.3 (92.7)
  IgA at 1 Year: number analyzed (Participants) | 23
  IgA at 1 Year | 111.6 (52.1)
  IgG at Baseline: number analyzed (Participants) | 30
  IgG at Baseline | 987.5 (343.2)
  IgG at 1 Year: number analyzed (Participants) | 23
  IgG at 1 Year | 1004 (521.9)
  IgM at Baseline | 102.8 (48.4)
  IgM at 1 Year: number analyzed (Participants) | 23
  IgM at 1 Year | 96 (85.2)

15. Secondary Outcome: Participants With Infections of Maximum Grade 2 and Grade 3
Description: Number of participants who reported the Maximum Infection Severity of Grade 2 and Grade 3. Only grade 2 and grade 3 infections occurring post transplantation were reported on the study. Grade 2 and grade 3 infections are defined by the BMT CTN Technical MOP. Higher infection grade indicates worse infection severity. The infection grading criteria are published online (https://bmtctn.net/administrative-manual-procedures-moppolicy-guidelines). Severity of grade 1, 2 and 3 are described for bacterial, fungal, viral, parasitic, and nonmicrobiological infections. For example, grade 2 fungal infections are defined as candida esophagitis, or proven or probably fungal sinusistis confirmed radiologically without orbital, brain or bone involvement. Grade 3 fungal infections are defined as Fungemia including candidemia, Proven or probably invasive fungal infections, Disseminated infections with histoplasmosis, blastomycosis, coccidiomycosis, or Cryptococcus, or Pneumocystis jiroveci pneumonia.
Time Frame: 1 Year
Population: Analysis Population includes transplanted participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
Participants
  None | 12
  Grade 2 | 12
  Grade 3 | 7

16. Secondary Outcome: Frequencies of Infections Categorized by Infection Type
Description: The number of systemic infections is reported. Infections are categorized by infection type. A participant can report multiple types of infections, so the categories are not mutually exclusive for participants. All grade 2 and grade 3 infections, as defined by the BMT CTN Technical MOP, occurring post transplantation were reported on the study.
Time Frame: 1 Year
Population: Analysis Population includes transplanted participants.
Measure: Number; unit: infections
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
infections
  Bacterial infection | 26
  Viral infection | 32
  Fungal infection | 3
  Protozoal infection | 0
  Other infection | 3

17. Secondary Outcome: Percentage of Participants With Cytomegalovirus (CMV), Epstein Barr Virus (EBV) or Post-Transplant Lymphoproliferative Disease (PTLD)
Description: CMV viremia and disease, EBV viremia, and PTLD are monitored and reported per protocol. The cumulative percentage of each outcome was estimated with a 95% confidence interval using the Aalen-Johansen estimator with death prior to event treated as a competing risk.
Time Frame: 1 Year
Population: Analysis Population includes transplanted participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
percentage of participants
  Cumulative Percentage of Participants with EBV | 9.7 [2.4 to 23.2]
  Cumulative Percentage of Participants with CMV | 22.6 [9.8 to 38.6]
  Cumulative Percentage of Participants with PTLD | 6.5 [1.1 to 18.9]

18. Secondary Outcome: Participants With Grade 3-5 Toxicities by SOC
Description: Toxicities are evaluated for the study participants at Day 28, Day 56, Day 100, Day 180 and Day 365 post-transplant and graded using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Grade 3-5 toxicities are reported with higher grade indicating worse outcomes. Toxicities are summarized here by system organ class (SOC). A participant can report multiple toxicities, so the categories are not mutually exclusive for participants.
Time Frame: 1 Year
Population: Analysis Population includes transplanted participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 31
Participants
  Abnormal Liver Symptoms | 7
  Blood and Lymphatic Disorders | 1
  Cardiovascular Disorders | 15
  Chemistry/Investigations | 2
  GI Disorders | 10
  General Disorders | 5
  Hemorrhagic Disorders | 3
  Hepatic Disorders | 6
  Immune System Disorders | 1
  Metabolism and Nutrition Disorders | 7
  Musculoskeletal and Connective Tissue Disorders | 1
  Nervous System Disorders | 4
  Renal Disorders | 5
  Respiratory, Thoracic and Mediastinal Disorders | 8
  Total (any of above SOC) | 23

19. Secondary Outcome: Health Related Quality of Life (HR-QoL) - Medical Outcomes Study Short Form (MOS SF-36)
Description: HR-QoL will be measured using patient reported surveys at baseline and then at Day 100, Day 180, and Day 365 post-transplant. The MOS SF-36 is used for adult participants (> 18 years). MOS SF-36 is a 36-item general assessment of HR-QoL with eight components: Physical Functioning, Role Physical, Pain Index, General Health Perceptions, Vitality, Social Functioning, Role Emotional, and Mental Health Index. Each domain is positively scored with higher scores associated with positive outcome. The scale is 0 to 100 where 0 is maximum disability and 100 is no disability. The Physical Component Summary (PCS) and Mental Component Summary (MCS) were used as the outcome measures in summarizing the SF-36 data for this study. These two summaries have the same score scale and Interpretation.
Time Frame: Baseline, Day 100, 6 Months, and 1 Year
Population: Analysis Population includes transplanted adult participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 18
score on a scale
  PCS at Baseline: number analyzed (Participants) | 15
  PCS at Baseline | 37.9 (7.9)
  PCS at Day 100: number analyzed (Participants) | 16
  PCS at Day 100 | 41.8 (11.6)
  PCS at 6 Months: number analyzed (Participants) | 16
  PCS at 6 Months | 44.3 (9.9)
  PCS at 1 Year: number analyzed (Participants) | 10
  PCS at 1 Year | 47.5 (8.1)
  PCS Change at Day 100 from baseline: number analyzed (Participants) | 14
  PCS Change at Day 100 from baseline | 4 (13.8)
  PCS Change at 6 Months from baseline: number analyzed (Participants) | 14
  PCS Change at 6 Months from baseline | 6.6 (11.6)
  PCS Change at 1 Year from baseline: number analyzed (Participants) | 9
  PCS Change at 1 Year from baseline | 10.4 (6.6)
  MCS at Baseline: number analyzed (Participants) | 15
  MCS at Baseline | 45.7 (13.2)
  MCS at Day 100: number analyzed (Participants) | 16
  MCS at Day 100 | 49.4 (14.2)
  MCS at 6 Months: number analyzed (Participants) | 16
  MCS at 6 Months | 50.4 (11.2)
  MCS at 1 Year: number analyzed (Participants) | 10
  MCS at 1 Year | 48.6 (14.9)
  MCS Change at Day 100 from baseline: number analyzed (Participants) | 14
  MCS Change at Day 100 from baseline | 4.8 (14)
  MCS Change at 6 Months from baseline: number analyzed (Participants) | 14
  MCS Change at 6 Months from baseline | 6 (10.2)
  MCS Change at 1 Year from baseline: number analyzed (Participants) | 9
  MCS Change at 1 Year from baseline | 2.2 (10.7)

20. Secondary Outcome: Health Related Quality of Life (HR-QoL) - PedsQL Stem Cell Transplant Module
Description: HR-QoL will be measured using patient reported surveys at baseline and then at Day 100, Day 180, and Day 365 post-transplant. The PedsQL Stem Cell Transplant Module for pediatric participants (8 years through 18 years). The PedsQL Stem Cell Transplant Module is a 46-item instrument that measures HR-QoL in children and adolescents undergoing hematopoietic stem cell transplant, and is developmentally appropriate for self-report in ages 8 through 18 years. The score ranges from 0 to 100 with higher scores associated with positive outcome.
Time Frame: Baseline, Day 100, 6 Months, and 1 Year
Population: Analysis Population includes transplanted pediatric participants. Four participants are under age 8 and not eligible for PedsQL assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Haplo Bone Marrow HSCT
Number analyzed (Participants) | 9
score on a scale
  PedsQL at Baseline | 72.8 (13.6)
  PedsQL at Day 100: number analyzed (Participants) | 7
  PedsQL at Day 100 | 86.5 (15.4)
  PedsQL at 6 Months: number analyzed (Participants) | 8
  PedsQL at 6 Months | 84.4 (12.5)
  PedsQL at 1 Year: number analyzed (Participants) | 6
  PedsQL at 1 Year | 93.3 (6.9)
  PedsQL Change at Day 100 from baseline: number analyzed (Participants) | 7
  PedsQL Change at Day 100 from baseline | 11.4 (16.2)
  PedsQL Change at 6 Months from baseline: number analyzed (Participants) | 8
  PedsQL Change at 6 Months from baseline | 9.5 (15.4)
  PedsQL Change at 1 Year from baseline: number analyzed (Participants) | 6
  PedsQL Change at 1 Year from baseline | 18.7 (11.1)

ADVERSE EVENTS:
Time Frame: Adverse event reporting and monitoring were conducted throughout the study, up to 1 year.
Description: An AE is any undesirable sign, symptom or medical condition or experience that develops or worsens after starting the first dose of study treatment or any procedure specified in the protocol, regardless of relationship to the study. A SAE is any AE that results in one of the followings, regardless of causality and expectedness: death, life-threatening, inpatient hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect, or an important medical event.
Groups:
- Enrolled Participants: Participants will be treated with a preparative regimen of Antithymocyte Globulin (ATG) (4.5 mg/kg), fludarabine (150 mg/m^2), cyclophosphamide (29 mg/kg), and low dose total body irradiation (TBI) (200 cGy) before undergoing the haplo HSCT. GVHD prophylaxis will be with post-HSCT cyclophosphamide (100 mg/kg), tacrolimus, and mycophenolate mofetil (MMF). G-CSF will be administered post-transplant.
Arm/Group | Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 7/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Participants (N=32)
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) — Incarcerated inguinal hernia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT02918292/Prot_SAP_ICF_000.pdf